CLINICAL TRIAL: NCT04838288
Title: Cognitive Outcomes and Quality of Life in Stable Renal Transplant Patients Switched FromTwice-Daily Tacrolimus to Envarsus XR™
Brief Title: Cognitive Outcomes in Stable Renal Transplant Patients Switched FromTacrolimus to Envarsus XR™
Acronym: OPERATOR
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Veloxis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Anthony Langone, Associate Professor, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201108
Record Dates: First submitted 2021-03-31; First posted 2021-04-09 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2024-08

CONDITIONS: Renal Transplant
Keywords: cognitive function; Quality of life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Change from Prograf to Envarsus (Experimental): All participants will be switched from Prograf to Envarsus
  Interventions: Drug: Change from Prograf to Envarsus XR

INTERVENTIONS:
Drug: Change from Prograf to Envarsus XR — Change from Tacrolimus taken twice a day to Envarsus XR taken once a day
  Other Names: Change from Tacrolimus to Envarsus XR

SUMMARY:
The purpose of this study is to assess cognitive outcome and quality of life in stable renal transplant patients treated with twice daily tacrolimus at baseline and after switching to Envarsus XL. The study is designed to see if switching patients from Tacrolimus to Envarsus treatment improves cognitive function.

DETAILED DESCRIPTION:
Patients with chronic kidney disease most commonly show cognitive impairments involving attention, memory, executive functions, and mental processing speed. Although data have demonstrated improvements in cognition following kidney transplant and the reversibility of the memory problems evidenced in dialysis, neurotoxicity in transplant patients occurs in >40-50% of the patients treated with tacrolimus. Attention and working memory impairment have been observed in patients treated with sirolimus or tacrolimus, while cyclosporine-treated patients demonstrated performance similar to that of healthy volunteer controls, which may indicate that the cognitive deficit found was partly related to treatment. ENVARSUS XR is a new FDA-approved formulation of tacrolimus. A hallmark difference between ENVARSUS XR and other forms of once- and twice-daily tacrolimus products is the unique, proprietary MeltDose® drug delivery technology (Veloxis Pharmaceuticals, Hørsholm, Denmark) which reduces tacrolimus' particle size to a molecular level. The decreased surface area of the drug particles results in complete absorption and increased bioavailability in a once-daily dosing formulation. In stable kidney transplant patients, ENVARSUS XR pharmacokinetics are characterized by a steadier and more consistent concentration time profile over 24 hours, reduced peak and peak-to-trough fluctuations and similar exposure while benefiting from ~ 20% less total daily dose than twice daily tacrolimus. This open-label, prospective phase clinical trial is designed to evaluate whether switching patients from TAC-IR to ENVARSUS XR treatment improves cognitive function.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be able to understand English and provide written informed consent;
2. Males and females between 18 and 70 years of age;
3. Recipients of a primary or secondary kidney transplant 4 weeks to 10 years prior to screening;
4. Patients receiving a stable dose (i.e., no dose adjustments) of TAC-IR for a minimum of 4-7 days at screening;
5. Patients with a screening TAC-IR trough level of 3-9 ng/mL, measured between Day -7 to 0;
6. Women of childbearing potential must have a negative urine pregnancy test at screening;
7. Patients must be willing to commit to and comply with the schedule of study visits.
8. The patient is not scheduled to begin any new medication that could interfere with tacrolimus blood levels, including prescription and over-the-counter medications, herbal or food supplements (including grapefruit and pomegranate products), or medications listed in Appendix 1.

Exclusion Criteria:

1. Recipients of any transplanted organ other than kidney;
2. Patients with an estimated glomerular filtration rate (eGFR) (MDRD4) < 25 mL/min at screening;
3. Patients with significant visual impairments affecting their ability to complete the study requirements and assessments: patient's vision is 20/200 or worse;
4. Patients with significant hearing impairments affecting their ability to complete the study requirements and assessments, based on Investigator discretion;
5. Patients with any severe medical condition (including infection) requiring acute or chronic treatment that in the Investigator's opinion would interfere with study participation;
6. Patients who have a history of any of the following, based on documentation of clinical conditions and concomitant medications in the medical records:

   * Cognitive decline secondary to stroke, per Investigator discretion
   * Dementia
   * Resected or existing brain tumor
   * Acute or chronic bipolar psychosis or schizophrenia per Investigator discretion
   * Mental retardation
   * Moderate or severe traumatic brain injury
   * Failure of any major organ other than the kidneys (e.g., end-stage liver disease)
   * Known non-adherence (defined as documentation in the patient chart of multiple missed visits and/or medication doses) which in the Investigator's opinion would interfere with the objectives of the study
7. Patients with medical history of hypertension or diabetes which is unmanageable by medically approved intervention (e.g., medication/diet) as assessed by the Investigator;
8. Patients with acute or chronic depression, corresponding to a score of ≥20 (corresponding to moderate depression) on the BDI-II at screening;
9. Patients who are taking any acute or chronic medications that may impact reaction time, memory, or sleep habits, based on Investigator discretion;
10. Patients on concurrent immunosuppression with MMF (CellCept) or MPS delayed release tablets (Myfortic), or generic versions of these medications, as per SOC, who have not been on stable doses (i.e., no dose adjustments or formulation change) for at least 4-7 days prior to screening;
11. Patients receiving prednisone or equivalent >10 mg/day;
12. Patients with an episode of biopsy-proven or suspected acute rejection that requires treatment within 3 months of screening;
13. Patients who are being actively treated for cancer (with the exception of non-invasive basal cell or cutaneous squamous cell carcinoma);
14. Patients known to be human immunodeficiency virus (HIV) positive;
15. Patients with any form of current drug or alcohol abuse as assessed by the Investigator;
16. Patients who were treated with any other investigational agent within 1 month prior to screening;
17. Pregnant or nursing women or women planning to become pregnant, where pregnancy is defined as a state of the female patient after conception and until the termination of gestation, confirmed by a positive urine laboratory test; women of child-bearing potential, defined as all women physiologically capable of becoming pregnant who are unwilling to use a defined SOC birth control method; UNLESS they are:

    * Women whose career, lifestyle, or sexual orientation preclude intercourse with a partner
    * Women whose partners have been sterilized by medically approved means

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-06-22 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in cognitive function-Global on RBANS | Baseline to month 4
  Measured by the Global Composite Score on the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS). Total score can range from 40 to 160. Low score indicates cognitive impairment.
Change in cognitive function-Global on Covid-19 telephone battery | Baseline to month 4
  Measured by the global composite score of the Covid-19 Telephone Battery, should that be the primary outcome battery that we employ due to COVID limitation. Total score can range from 40 to 160. Low score indicates cognitive impairment.

SECONDARY OUTCOMES:
Change in cognitive function on Trail making part A | Baseline to month 4
  Measured by Trail making Part A. Maximum time given for TMT A is 150 seconds. Results are reported as the number of seconds required to complete the task; therefore, higher scores reveal greater impairment.
Change in cognitive function on Trail making part B | Baseline to month 4
  Measured by Trail making Part B. Maximum time given for TMT B is 300 seconds. Results are reported as the number of seconds required to complete the task; therefore, higher scores reveal greater impairment.
Change in quality of life | Baseline to Month 4
  Change in quality of life measured by WHODAS. The total score of WHODAS is the sum of all the 12 sub-scores and ranges from 0 to 48, with lower scores indicating better functioning. Total scores of 1-4 belong to mild disability, 5-9 to moderate disability, and 10-48 to severe disability
Impression of Improvement by PGI | baseline to month 4
  measured by PGI-I (Patient's Global Impression of Improvement). The PGI-I measures change since initiating a medication and is assessed on a 7-point Likert-type scale ranging from very much better (1) to very much worse (7)
Impression of Improvement by CGI | baseline to month 4
  measured by CGI-I (Clinical Global Impression of Improvement). The CGI-I measures change since initiating a medication and is assessed on a 7-point Likert-type scale ranging from very much improved (1) to very much worse (7).
Change of quality of sleep | Baseline to month 4
  measured by PIRS-20 (Pittsburgh Insomnia Rating Scale). The PIRS-20 total score is the sum of all items and ranges from 0 (good sleep) to 60 (bad sleep).3

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Langone, MD, Principal Investigator — VUMC
Locations (1):
- VUMC, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No